CLINICAL TRIAL: NCT03133195
Title: A Phase III, Randomized, Double Blind, Placebo Controlled Study to Evaluate the Effect of Teriparatide on Bone Union in Unstable Intertrochanteric Fracture Patients Treated With Proximal Femoral Nail Antirotation (PFNA)
Brief Title: The Effect of Teriparatide on Bone Union in Unstable Intertrochanteric Fracture Patients Treated With PFNA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: King Chulalongkorn Memorial Hospital (Other)
Responsible Party: Principal Investigator, Prof.Dr.Aree Tanavalee, M.D., Prof. Dr., M.D., King Chulalongkorn Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ORTHCU-2017-01
Record Dates: First submitted 2017-04-21; First posted 2017-04-28 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Unstable Intertrochanteric Fracture; Pertrochanteric Fracture of Femur, Closed
Keywords: Terriparatide, bone fracture healing, PFNA
MeSH Terms: interventions — Teriparatide; Vitamin D

STUDY DESIGN:
Intervention Model Description: The patients will be randomized in 1:1 ratio to receive Teriparatide or placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double blind, placebo-controlled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Teriparatide (Experimental): Teriparatide 20 μg subcutaneous once daily for 12 weeks
  Interventions: Drug: Teriparatide; Dietary Supplement: Calcium supplement; Dietary Supplement: Vitamin D
- Placebo (Placebo Comparator): Placebo subcutaneous once daily for 12 weeks
  Interventions: Drug: Placebo; Dietary Supplement: Calcium supplement; Dietary Supplement: Vitamin D

INTERVENTIONS:
Drug: Teriparatide — Teriparatide 20 μg subcutaneous once daily for 12 weeks (Patient self administration at home by pen injector)
  Other Names: r-Human parathyroid hormone
  Arms: Teriparatide
Drug: Placebo — Placebo subcutaneous once daily for 12 weeks. (Patient self administration at home by pen injector)
  Arms: Placebo
Dietary Supplement: Calcium supplement — 1000 mg/day of elemental calcium
Dietary Supplement: Vitamin D — 20,000 IU/week of vitamin D2

SUMMARY:
Phase III, prospective, randomized, parallel, double blind, placebo-controlled study to determine whether Teriparatide can accelerate bone healing in unstable intertrochanteric fracture patients treated with Proximal Femoral Nail Antirotation (PFNA) assessed by radiographic and clinical outcomes.

DETAILED DESCRIPTION:
Patients will undergo screening assessment to determine the eligibility for study participation and will be randomized in 1:1 ratio to receive Teriparatide 20 μg or placebo subcutaneous once daily for 12 weeks.

All patients will receive supplements of 1000 mg/day of elemental calcium and 20,000 IU/week of vitamin D2.

Patients will be scheduled to clinic visit for radiographic and clinical assessment at 2, 6,12 and 24 weeks postoperatively. Each participant will be in the study for 6 months in total.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patient, age ≥ 50 years at the time of screening
2. Unstable intertrochanteric fracture (AO/OTA 31-A2 and 31-A3)
3. Treated by proximal femoral nail antirotation (PFNA)

Exclusion Criteria:

1. Known hypersentivity to teriparatide or any form of PTH or analogue
2. Metabolic bone disease other than primary osteoporosis (including Hyper Parathyroidism and Paget's disease of bone)
3. Increased baseline risk of osteosarcoma (Paget's disease of the bone, previous primary skeletal malignancy, or skeletal exposure to therapeutic irradiation)
4. History of malignant neoplasm in the 5 years prior to the study (with the exception of superficial basal cell carcinoma or squamous cell carcinoma) and carcinoma in situ of the uterine cervix treated less than 1 year prior to the study.
5. Pre-existing of hypercalcemia (total serum calcium >10.5 mg/dL or 2.6 mmol/L)
6. Abnormally elevated serum intact parathyroid hormone at screening (serum PTH > 70 pg/mL)
7. Severe vitamin D deficiency (25-hydroxyvitamin D < 12 ng/mL)
8. Unexplained elevations of alkaline phosphatase (ALP > 120 UL)
9. Severe renal impairment (CrCL < 30 mL/min)
10. Current treatment with digoxin and necessary to continue use during the study
11. Concurrent treatment with oral bisphosphonates, selective estrogen receptor modulator (SERMs), calcitonin, estrogen (oral, transdermal, or injection), progestin, estrogen analog, estrogen agonist, estrogen antagonist or tibolone, and active vitamin D3 analogs. (Previous treatment is allowed but must be discontinued at screening)
12. Previous treatment with strontium ranelate for any duration, intravenous bisphophonates within 12 months prior to the screening date, and/or denosumab within 6 months prior to the screening.
13. Previous treatment with teriparatide, PTH or other PTH analogs, or prior participation in any other clinical trial studying teriparatide, PTH or other PTH analogs

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-05-17 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
Time to healing assessed by radiographic evidence | from randomization, assessed up to 24 months
  Fracture is judged to be healed radiographically if bridging callus was evident on 3 of 4 cortices as seen on two views (cortical bridging of three cortices)

SECONDARY OUTCOMES:
Clinical evidence of healing assessed by Harris Hip Score as one of functional outcomes | from randomization, assessed up to 24 months
  Harris Hip Score (90-100: Excellent, 80-89: Good, 70-79: Fair, <70 poor)
Clinical evidence of healing assessed by weight bearing ability as one of functional outcomes | from randomization, assessed up to 24 months
  Weight bearing ability (Non weight bearing, Partial weight bearing, Full weight bearing)
Clinical evidence of healing assessed by walking ability as one of functional outcomes | from randomization, assessed up to 24 months
  Walking ability (Independent walking, Assisted walking, Bedridden)

CONTACTS AND LOCATIONS:
Overall Officials: Prof.Dr.Aree Tanavalee, M.D., Principal Investigator — Chulalongkorn University
Locations (1):
- Faculty of Medicine Chulalongkorn University, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Undecided